CLINICAL TRIAL: NCT02908568
Title: Effect of Stimulation of the Proprioceptive Trigeminocardiac Reflex Through Medical Device for the Pain of Patients With Temporomandibular Disorders
Brief Title: Stimulation of the Proprioceptive Trigeminocardiac Reflex
Acronym: PTCRSTIM
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azienda USL 12 Versilia (Other)
Responsible Party: Principal Investigator, PROF. UGO COVANI, Azienda USL 12 Versilia, Azienda USL 12 Versilia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ISTITUTO STOMATOLOGICO TOSCANO
Record Dates: First submitted 2016-09-07; First posted 2016-09-21 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Temporomandibular Joint Disorders
Keywords: mandibular stretching, trigeminocardiac reflex
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Spring device (Experimental): Brisk dilatation of fhe mouth.
  Interventions: Device: Spring device
- Mandible stimulator (Sham Comparator): Stimulation of fhe mouth.
  Interventions: Device: Mandible stimulator

INTERVENTIONS:
Device: Spring device — Brisk dilatation of fhe mouth.
  Arms: Spring device
Device: Mandible stimulator — Stimulation of fhe mouth.
  Arms: Mandible stimulator

SUMMARY:
Study over muscular stretching to reduce pain the oral cavity.

DETAILED DESCRIPTION:
It is a current opinion that muscular stretching is able to reduce pain and to allow increase of the opening excursion at the joints. To investigate this possibility in the face, the investigators developed a method of stretching associated with large dynamic jaws during chewing using a special device (Spring Device ®) for ten minutes, allowing the muscles of the oral cavity to relax. The height of the bite was set as two-thirds of the maximum opening (max. 2 cm.) of the mouth at rest (without forcing) thus avoiding maintaining the head of the condyle at maximum aperture for a long time. The subjects were then analyzed by means of kinesiography to determine the changes in the vertical dimension. Increasing stretching produces neuromuscular relaxation and a reduction of pain. This study showed that this therapy induces oral and extraoral pain reduction and increases neck mobility and mouth opening. The stimulation of trigeminal receptors is an important drive for therapy in the trigeminocardiac reflex (TCR).

ELIGIBILITY:
Inclusion Criteria:

* All the subjets up to seventy years

Exclusion Criteria:

* Subjects under eight years

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Mandibular stretching influences the temporomandibular disorders | up to 24 weeks
  It is a current opinion that muscular stretching is able to reduce pain and to allow increase of the opening excursion at the joints.
  To investigate this possibility in the face, the investigators developed a method of stretching associated with large dynamic jaws during chewing using a special device (Spring Device ®) for ten minutes, allowing the muscles of the oral cavity to relax.

SECONDARY OUTCOMES:
mandibular stretching induces a reduction of facial contraction and decrease of heart rate | up to 24 weeks
  Those effects are described as trigemino-cardiac reflex. Application of a spring device (which consists of thin sheet of surgical steel bent in to a loop) induces a decrease of blood pressure and heart rate.

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Tonlorenzi D, Brunelli M, Conti M, Covani U, Traina G. An observational study of the effects of using an high oral splint on pain control. Arch Ital Biol. 2019 Sep 30;157(2-3):66-75. doi: 10.12871/00039829201923. PMID 31821530